CLINICAL TRIAL: NCT01888900
Title: Unraveling the Mechanisms of Non-Response in Patients With and Without Cirrhosis Due to Chronic Hepatitis C
Brief Title: New Treatment Response in People With and Without Cirrhosis From Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130150; 13-DK-0150; 13-DK-0150 (Other: National Institutes of Health)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Cirrhosis; Chronic Hepatitis C; Hepatitis C; Hepatitis C, Chronic
Keywords: Hepatitis C; Non-Responders; Direct Acting Antivirals; Interferon Free; Cirrhosis
MeSH Terms: conditions — Fibrosis; Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatitis C Virus Genotype 1A with QUAD (Experimental): Subjects will be started on combination therapy with asunaprevir, daclatasvir, peginterferon alfa-2a and ribavirin for 24 weeks.
  Interventions: Drug: QUAD
- Hepatitis C Virus Genotype 1B with DUAL (Experimental): Subjects will receive combination therapy with asunaprevir and daclatasvir alone for 24 weeks and undergo paired liver biopsies, pre-treatment and either at 2 or 4 weeks after starting therapy.
  Interventions: Drug: DUAL

INTERVENTIONS:
Drug: DUAL — Asunaprevir and Daclatsvir
  Arms: Hepatitis C Virus Genotype 1B with DUAL
Drug: QUAD — Asunaprevir, daclatsvir, peginterferon and ribavirin
  Arms: Hepatitis C Virus Genotype 1A with QUAD

SUMMARY:
Background:

- Some people who have chronic hepatitis C do not respond to the usual treatment with peginterferon and ribavirin. New chronic hepatitis treatments are being developed that may work better for different people. The treatments will look at how specific genes interact with the drugs. Researchers want to see how well these new drugs work in people whose chronic hepatitis C has not responded or only partly responded to the usual treatment drugs.

Objectives:

- To compare new treatments for people with chronic hepatitis C.

Eligibility:

- Individuals at least 18 years of age who have chronic hepatitis C that has not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Liver scans and a biopsy will be taken before the start of treatment.
* Participants will be separated into two groups. One group will have the new treatment drugs (assunaprevir and daclatasvir). The second group will have these two drugs as well as peginterferon and ribavirin. All participants will have an initial 4-day hospital stay with regular blood tests to see how the start of the treatment works.
* The first group will take the new study drug tablets daily for 24 weeks. Those who do not respond to this treatment will also start to take peginterferon and ribavirin, and the treatment will continue for 24 weeks after starting the additional drugs.
* The second group will take all four drugs according to the standard dosing schedule for 24 weeks.
* Treatment will be monitored with frequent blood tests. Liver scans, biopsies, and other tests will be performed as directed by the study doctors.
* Participants will have 24 weeks of regular followup visits.

DETAILED DESCRIPTION:
Up to 70 patients with chronic hepatitis C, genotype 1, who were partial or null responders to optimal therapy with the combination of peginterferon and ribavirin will be enrolled into this pilot study on the use of asunaprevir and daclatasvir together or in combination with peginterferon alfa-2a and ribavirin to improve response to antiviral therapy. Two separate studies will be conducted based upon HCV genotype 1 subtype. For patients with HCV genotype 1b: Will undergo baseline testing for NS5A RAVs known to confer resistance to daclatasvir (L31/Y93). Subjects who harbor these NS5A resistance associated variants will be excluded from receiving dual therapy but would be offered quad therapy and managed as a HCV genotype 1a subject. After medical evaluation and liver biopsy, 30 HCV genotype 1b patients will receive combination therapy with asunaprevir and daclatasvir alone for 24 weeks and undergo paired liver biopsies, pre-treatment and either at 2 or 4 weeks after starting therapy. Patients in whom HCV RNA is greater than or equal to LLOQ at 8 weeks will either discontinue therapy at that point (early stopping rule for futility) or may have rescue therapy instituted at the discretion of the investigator with a QUAD regimen (asunaprevir and daclatasvir plus peginterferon and ribavirin) provided they meet pre-specified inclusion criteria. For patients with HCV genotype 1a: After medical evaluation and liver biopsy 40 (15 with cirrhosis and 15 with Ishak fibrosis 0-2; the remaining 10 slots will be allocated for individuals who do not meet the histological entry requirement i.e. Ishak 3-4) HCV genotype 1a patients will be started on combination therapy with asunaprevir, daclatasvir, peginterferon alfa-2a and ribavirin for 24 weeks. Patients will be randomized to undergo a second liver biopsy at study week 4 after starting therapy either before or 6 hours after the next scheduled peginterferon dose to assess intrahepatic interferon stimulated gene expression. Intrahepatic drug concentrations of asunaprevir and daclatasvir will be measured as part of an ancillary study. Patients in whom HCV RNA is greater than or euqal to LLOQ at 8 weeks will discontinue therapy (early stopping rule for futility). Routine serum chemistries, complete blood counts and HCV RNA levels will be monitored more frequently for the initial 4 days and then at standard intervals during the period of antiviral therapy. The major endpoints will be changes in interferon stimulated gene and protein expression in the liver and changes in HCV RNA levels in liver and serum between baseline and 4 weeks. Secondary endpoints will be rates of sustained virologic response 12 and 24 weeks off therapy.

ELIGIBILITY:
-INCLUSION CRITERIA:

INCLUSION CRITERIA FOR BOTH GENOTYPES 1a and 1b:

1. Adults, ages 18 and above
2. Chronic hepatitis C (HCV RNA in serum for more than 6 months)
3. HCV Genotype 1
4. HCV RNA in serum above 10,000 IU/mL
5. Non-response to previous therapy with peginterferon and ribavirin categorized as null-response as defined by a less than 1 log IU/mL decline in HCV RNA at treatment week 4 or a less than 2 log IU/mL decline in HCV RNA at treatment week 12; and partial response as defined by a greater than or equal to 2 log decrease in HCV RNA at treatment week 12 but continued detection of HCV RNA at treatment week 24
6. No contraindications to agents being used (asunaprevir, daclatasvir, peginterferon and ribavirin).
7. No evidence or history of hepatic decompensation.
8. Females of childbearing potential must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours before the first dose of study drug.
9. Women of childbearing potential (WOCBP) and men must use highly effective methods of birth control to minimize the risk of pregnancy. WOCBP must follow instructions for birth control for the entire duration of the study including a minimum of 24 weeks after the last dose of P/R. Birth control requirements are or WOCBP and men who are sexually active with WOCBP
10. Women must not be breastfeeding
11. Fully informed, written consent to the study including repeat liver biopsy.

ADDITIONAL INCLUSION CRITERIA FOR GENOTYPE 1a

1) Liver biopsy showing Ishak stages 0-2 or 5-6 within 12 weeks of initiating therapy OR a prior biopsy performed within 96 weeks of screening visit WITH saved tissue. Up to 10 subjects who do not fulfill the entry histologic criteria will be allowed to participate in the trial at the discretion of the investigator.

ADDITIONAL INCLUSION CRITERIA FOR GENOTYPE 1b

1. Baseline sequence analysis of the NS5A region to exclude presence of mutations known to confer resistance to daclatasvir.

INCLUSION CRITERIA FOR GT 1b SUBJECTS WHO RECEIVE RESCUE THERAPY AT THE DISCREATION OF THE INVESTIGATOR (THESE CRITERIA MUST BE ASSESSED PRIOR TO INITIATIONOF PEG INFa/RBV THERAPY):

Important: In addition to the Inclusion Criteria listed above, the following

Inclusion Criteria apply to all Rescue Subjects:

a) Subject met a definition of virologic breakthrough or treatment futility, defined

as:

i) Any confirmed > 1 log10 increase in HCV RNA from nadir, OR;

ii) Any confirmed HCV RNA greater than or equal to Lower Limit of quantification (LLOQ) after confirmed HCV RNA <LLOQ Target Not Detected while on treatment, OR;

iii) Any confirmed HCV RNA greater than or equal to LLOQ at Week 8. Measurements should be confirmed within 2 weeks of the Week 8 result;

b) HCV RNA < 400,000 IU/mL at the last assessment; This cut-off was chosen because it is felt that peginterferon and ribavirin would be ineffective at higher viral loads in prior non-responders to peginterferon and ribavirin with viral breakthrough.

c) Women of childbearing potential (WOCBP)1 and men must use highly effective methods of birth control to minimize the risk of pregnancy. WOCBP must follow instructions for birth control for the entire duration of the study including a minimum of 24 weeks after the last dose of P/R. Birth control requirements are or WOCBP (see Section C.5 for the definition of WOCBP) and men who are sexually active with WOCBP;

i) Two (2) forms of birth control are required from time of screening throughout the duration of the on-treatment study period and for at least 24 weeks after the last dose of RBV (or the duration specified by the country-specific RBV label, whichever is longer), in such a manner that the risk of pregnancy is minimized. Examples of highly effective birth control include:

-condom with spermicide;

-diaphragm and spermacide;

-cervical cap and spermacide

* female condom;
* intrauterine devices (IUDs);

Oral contraceptive pills (OCPs) may be used in this study but cannot be considered as an effective form of contraception for WOCBP subjects.

ii) Exceptions include:

1. WOCBP who are not heterosexually active or who have male partners who have been vasectomized for a minimum of 6 months with a history of confirmed azoospermia;
2. Sexually active men who are vasectomized for a minimum of 6 months with a history of confirmed azoospermia.

   d) WOCBP must have a negative serum or urine pregnancy test [minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)] within 24 hours prior to the start of P/R. Female subjects must agree to the pregnancy testing requirements of this protocol;

   e) Women must not be breastfeeding;

   f) Male Subjects: Requirements (based on RBV label):

   i) Male subjects (unless vasectomized for at least 6 months with a history of confirmed azoospermia) with female partners who are WOCBP must agree to inform their female partners of the protocol-specified effective birth control methods requirement and pregnancy testing recommendations during treatment and post-treatment (i.e., two forms of effective methods of birth control and monthly pregnancy testing while the subject is enrolled in the study and 6 months following discontinuation of RBV [or for the post-treatment duration specified in the country-specific RBV label]), and agree to adhere to these recommendations both on-treatment and during the post-treatment follow-up period;

ii) Male subjects must confirm that their female sexual partners are not pregnant at the time of screening.

EXCLUSION CRITERIA:

Exclusion Criteria for Genotypes 1b:

1. Medical History and Concurrent Diseases

   1. Liver or any other organ transplant (including hematopoietic stem cell transplants) other than cornea and hair;
   2. Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment
   3. Documented or suspected HCC, as evidenced by previously obtained imaging studies or liver biopsy (or on a screening imaging study/liver biopsy if this was performed)
   4. Evidence of decompensated liver disease including, but not limited to, radiologic criteria, a history or presence of ascites, bleeding varices, or hepatic encephalopathy
   5. Evidence of a medical condition contributing to chronic liver disease other than HCV (such as, but not limited to: hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
   6. History of chronic hepatitis B virus (HBV) as documented by HBV serologies (eg, HBsAg-seropositive). Subjects with resolved HBV infection may participate (eg, HBsAb-seropositive with concurrent HBsAg-seronegative)
   7. Any gastrointestinal disease or surgical procedure that may impact the absorption of study drug. (Subjects who have had cholecystectomy are permitted to enter the study)
   8. History of HIV infection
   9. Hemophilia
   10. Uncontrolled diabetes (any subject with a confirmed screening HgA1c greater than or equal to 8.5 must be excluded)
   11. Confirmed, uncontrolled hypertension (any screening systolic blood pressure greater than or equal to 160 mmHg or diastolic blood pressure greater than or equal to 100 mmHg should be excluded unless discussed with the central medical monitor)
   12. Any other medical and/or social reason, including active substance abuse as defined by DSM-IV, Diagnostic Criteria for Drug and Alcohol Abuse, which in the opinion of the investigator would make the candidate inappropriate for participation in this study
   13. History of severe psychiatric disorders including but not limited to, schizophrenia, psychosis, bipolar disorder, post-traumatic stress disorder, mania, etc.
   14. Inability to tolerate oral medication;
   15. Poor venous access

       2. Physical and Laboratory Test Findings

Note: Growth factors must not be used to achieve eligibility criteria.

1. ALT greater than or equal to 10 times ULN
2. Total bilirubin greater than or equal to 34 micromoles per liter (greater than or equal to 2 mg/dL) unless the subject has documented history of Gilbert s disease
3. Albumin < 3.5 g/dL (35 g/L)
4. Creatinine clearance (CrCl) less than or equal to 50 ml/min (as estimated by Cockcroft and Gault)
5. Platelets < 50 times 10(9) cells/L
6. ANC < 0.5 times 10(9) cells/L
7. Hemoglobin < 8.5 g/dL
8. INR greater than or equal to 1.7
9. Alpha-fetoprotein (AFP):

i) AFP > 100 ng/mL OR

ii) AFP greater than or equal to 50 ng/mL and less than or equal 100 ng/mL requires a liver ultrasound and subjects with findings suspicious for HCC are excluded

j) QTcF or QTcB > 500 msec

3. Allergies and Adverse Drug Reaction

a) History of hypersensitivity to drugs with a similar biochemical structure to asunaprevir

or daclatasvir.

4. Prohibited Treatments and /or Therapies

1. Exposure to any investigational drug or placebo within 4 weeks of study drug administration;
2. Prior exposure to any HCV DAA;
3. Prior exposure to pegIFN or RBV within 12 weeks prior to screening;
4. Subjects receiving all tricyclic anti-depressants (TCAs) including amitriptyline, clomipramine, desiprmine, dosepin, imipramine, nortriptyline, protriptyline; OR selective serotonin reuptake inhibitors (SSRIs) including fluoxetine, fluvoxamine, paroxetine and

sertraline; OR additional agents including venlafaxine, duloxetine, aripiprazole and mirtazapine within 2 weeks prior to Day 1; (subjects may switch to non-prohibited antidepressant therapies (eg citalopram, escitalopram and bupropion) within 2 weeks prior to

Day 1). The study eligibility of subjects on any anti-depressant not listed above, may be considered after a consultation with the central medical monitor, prior to Day 1;

5. Sex and Reproductive Status

1. Sexually active men whose partners are pregnant at screening are excluded from this study

   6. OTHER EXCLUSION CRITERIA

a) Prisoners or subjects who are involuntarily incarcerated

b) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

C.5 Exclusion Criteria for Gt 1a subjects and 1b subjects who receive rescue therapy at discretion of the investigator (Prior to initiation of PegIFN /ribavirin therapy):

Important: In addition to the Exclusion Criteria listed above WITH THE EXCEPTION OF THE LABORATORY TESTS INDICATED IN SECTION C.4.2 A-H, the following

Exclusion Criteria apply to all Gt 1a and rescue subjects:

a) Severe psychiatric disease that would prohibit use of peg-IFN -2a as judged by the investigator including but not limited to:

i) Moderate or severe depression; Beck Depression Score greater than or equal to 15 during screening

ii) History of depression associated with hospitalized for depression,

electroconvulsive therapy, or depression resulting in a prolonged absence from work and/or significant disruptions from daily functions;

iii) Suicidal or homicidal ideation and/or attempt;

iv) History of severe psychiatric disorders including but not limited to,

schizophrenia, psychosis, bipolar disorder, post-traumatic stress disorder, mania, etc.;

b) History of hemoglobinopathies (e.g., thalassemia major or sickle cell anemia), diagnoses associated with an increased baseline risk for anemia (e.g., spherocytosis), hemolytic anemia, or diseases in which anemia would be medically problematic, or hemophilia;

c) Pre-existing ophthalmologic disorders considered clinically significant on eye exam, including retinal, examination. Note: all subjects with a history of diabetes or hypertension must have a documented eye exam within 12 months prior to initiation of P/R;

d) Thyroid-stimulating hormone (TSH) < 0.8 times LLN or > 1.2 times ULN of the laboratory reference range, unless

i) The subject is clinically euthyroid as determined by the investigator, AND

ii) Free T4 is greater than or equal to 0.8 times LLN and less than or equal to 1.2 times ULN

e) History of chronic pulmonary disease associated with functional limitation such as clinically significant chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidois, etc;

f) History of cardiomyopathy, coronary artery disease (including angina), interventional procedure for coronary artery disease (including angioplasty, stent procedure, or cardiac bypass surgery), ventricular arrhythmia, congestive heart failure, pulmonary hypertension, cardiomyopathy, or other clinically significant cardiac disease;

g) Historical or current ECG findings indicative of cardiovascular instability, including but not limited to evidence of significant myocardial ischemia, unstable re-entry phenomena, other significant dysarrhythmias and/or uncontrolled hypertension;

h) Immunologically-mediated disease (eg, inflammatory bowel disease [Crohn s disease, ulcerative colitis], celiac disease, rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma,

sarcoidosis, severe psoriasis requiring oral or injected treatment, or symptomatic thyroid disorder).

i) Any known contraindication to peg-IFN -2a or ribavirin, not otherwise specified.

j) Alanine aminotransferase (ALT) greater than 10 times ULN;

k) Total Bilirubin greater than or equal to 34 mol/L (greater than or equal to 2 mg/dL), unless subject has a documented history of Gilbert s disease;

l) INR greater than or equal to 1.7;

m) Albumin < 3.5 g/dL (35 g/L);

n) Platelets < 70 times 10(9) cells/L;

o) ANC < 1,500 cells/mm3 (confirmed ANC < 1,200 cells/mm3 for Black/African-Americans);

p) Hemoglobin < 12 g/dL (120 g/L) for women and < 13 g/dL (130 g/L) for men;

q) Creatinine Clearance (CrCl) less than or equal to 50 mL/min (as estimated by Cockcroft and Gault);

r) History of hypersensitivity to drugs with similar biochemical structure to pegIFN alpha or ribavirin

s) QTcF or QTcB > 500 msec;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patients will have serum stored from selected time points during this study. These specimens will be used for repeat virological testing and special tests as needed (such as for viral levels, HCV RNA sequencing, HCV resistance testing or measurement of serum levels of cytokines, IL28b testing or interferon induced genes) and for future research.

REFERENCES:
- [Background] Shepard CW, Finelli L, Alter MJ. Global epidemiology of hepatitis C virus infection. Lancet Infect Dis. 2005 Sep;5(9):558-67. doi: 10.1016/S1473-3099(05)70216-4. PMID 16122679
- [Background] Lavanchy D. The global burden of hepatitis C. Liver Int. 2009 Jan;29 Suppl 1:74-81. doi: 10.1111/j.1478-3231.2008.01934.x. PMID 19207969
- [Background] Esteban JI, Sauleda S, Quer J. The changing epidemiology of hepatitis C virus infection in Europe. J Hepatol. 2008 Jan;48(1):148-62. doi: 10.1016/j.jhep.2007.07.033. Epub 2007 Nov 5. PMID 18022726
- [Derived] Serti E, Park H, Keane M, O'Keefe AC, Rivera E, Liang TJ, Ghany M, Rehermann B. Rapid decrease in hepatitis C viremia by direct acting antivirals improves the natural killer cell response to IFNalpha. Gut. 2017 Apr;66(4):724-735. doi: 10.1136/gutjnl-2015-310033. Epub 2016 Jan 4. PMID 26733671
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0150.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatitis C Virus Genotype 1A: Subjects will be started on combination therapy with asunaprevir, daclatasvir, peginterferon alfa-2a and ribavirin for 24 weeks.
- Hepatitis C Virus Genotype 1B: Subjects will receive combination therapy with asunaprevir and daclatasvir alone for 24 weeks.
Period: Overall Study
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Started | 22 | 13
Completed (2 failures were switched from DUAL treatment to QUAD treatment.) | 22 | 11
Not Completed | 0 | 2
Not completed — failed treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Hepatitis C Virus Genotype 1B: Patients will receive combination therapy with asunaprevir and daclatasvir alone for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.50 (7.65) | 59.31 (11.06) | 57.54 (9.01)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 17 | 7 | 24
ALT [Mean (Standard Deviation); unit: U/L] — alanine aminotransferase
  U/L | 99.36 (52.84) | 78.08 (42.18) | 91.46 (49.68)
HCV RNA level [Mean (Standard Deviation); unit: log10(IU/ml)] — log with base 10 transformed HCV RNA
  log10(IU/ml) | 6.67 (0.49) | 6.72 (0.37) | 6.69 (0.44)
Race [Number; unit: participants]
  Asian | 1 | 2 | 3
  Black | 9 | 4 | 13
  White | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Changes in Interferon Stimulated Genes in the Liver
Description: Change in raw expression in interferon stimulated genes at week 2 or 4 compared to baseline is obtained by subtracting either 2 or 4 week measurement from baseline measurement. Negative values reflect a decrease in expression and positive values reflect an increase in expression.
  The raw gene expression data was normalized using quantile normalization based on all the genes in the microarray.
Time Frame: baseline and either 2 or 4 weeks
Population: one patient in genotype 1A arm was not included in primary outcome data collection due to late enrollment.
Measure: Median (Inter-Quartile Range); unit: relative expression
Groups:
- Hepatitis C Virus Genotype 1A: Patients will be started on combination therapy with asunaprevir, daclatasvir, peginterferon alfa-2a and ribavirin for 24 weeks.
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 21 | 11
relative expression
  ACADSB | -0.04915 [-0.20904 to 0.12412] | -0.35948 [-0.65364 to -0.32862]
  ACSM3 | -0.49980 [-0.64301 to -0.07697] | -0.79328 [-0.91284 to -0.47427]
  ADH6 | -0.11373 [-0.38039 to 0.03311] | -0.36659 [-0.73021 to -0.13545]
  ANXA9 | -0.07636 [-0.29628 to 0.03123] | -0.50104 [-0.66928 to -0.38972]
  APOA5 | -0.12453 [-0.45306 to 0.28019] | -0.48167 [-0.72870 to -0.29107]
  APOF | -0.26305 [-0.63316 to -0.06705] | -0.39732 [-0.95115 to -0.21099]
  BDH1 | -0.08100 [-0.29314 to 0.06585] | -0.27664 [-0.49475 to -0.12647]
  CCL19 | 0.61221 [-0.08379 to 1.13362] | 1.08586 [-0.62653 to 1.49427]
  CCL2 | 0.15200 [-0.15355 to 0.50558] | 0.66422 [0.43410 to 1.70929]
  CCL20 | 0.41719 [0.13460 to 0.78103] | 0.91927 [-0.01334 to 1.13015]
  CCL4 | 0.68293 [0.31016 to 1.13638] | 0.89852 [0.21807 to 1.07382]
  CXCL10 | 2.08246 [1.73241 to 2.57419] | 2.34623 [1.71264 to 2.91674]
  CXCL11 | 1.34781 [0.94627 to 1.89192] | 1.62034 [1.43302 to 1.92497]
  CXCL9 | 1.46361 [0.87882 to 2.60228] | 1.16119 [0.89738 to 1.92419]
  CYP1A1 | 0.31399 [-0.48087 to 1.25841] | -0.71461 [-1.34260 to -0.42217]
  CYP4A11 | -0.09207 [-0.37379 to 0.00367] | -0.21412 [-0.34514 to 0.03285]
  DDX58 | -0.11579 [-0.46440 to -0.00993] | 0.71105 [0.34121 to 1.41336]
  DDX60 | 0.15820 [0.06634 to 0.51348] | 1.75573 [1.38395 to 2.15565]
  EIF2AK2 | -0.30273 [-0.58088 to -0.13209] | 0.79761 [0.39253 to 1.08915]
  FDPS | 0.13720 [-0.31418 to 0.30542] | -0.62267 [-0.97700 to -0.23584]
  HMGCS2 | -0.12509 [-0.18190 to 0.00777] | -0.24445 [-0.41498 to -0.01065]
  IFI27 | -0.02793 [-0.14563 to 0.14139] | 0.95729 [0.74599 to 1.45239]
  IFI44L | -0.74607 [-1.12864 to -0.33525] | 2.33014 [0.88173 to 2.89601]
  IFI6 | 0.35068 [-0.09436 to 0.57536] | 0.44506 [-0.03475 to 1.32183]
  IFIH1 | -0.04591 [-0.25975 to 0.24874] | 1.11512 [0.86720 to 1.52474]
  IFIT1 | -0.07569 [-0.41657 to 0.30933] | 1.49718 [0.63654 to 2.04239]
  IFIT2 | 0.36377 [-0.18331 to 0.96812] | 1.09749 [0.14450 to 1.56788]
  IFIT3 | -0.00220 [-0.31494 to 0.34534] | 1.45782 [0.12098 to 1.92258]
  IFITM1 | 0.00657 [-0.13774 to 0.15923] | 0.87242 [0.52497 to 1.00591]
  IRF9 | -0.07023 [-0.23137 to 0.30435] | 0.07203 [-0.43579 to 0.44433]
  ISG15 | 0.25402 [-0.02712 to 0.37972] | 2.25228 [1.67411 to 2.57665]
  ISG20 | 0.55260 [0.11923 to 0.77920] | 0.79333 [0.17554 to 1.01774]
  LCAT | -0.23342 [-0.42605 to -0.13411] | -0.28993 [-0.61976 to -0.10027]
  LIPC | -0.16928 [-0.47942 to -0.00974] | -0.77129 [-1.09584 to -0.32804]
  LSS | 0.04955 [-0.33891 to 0.32346] | -0.87048 [-1.06593 to -0.28066]
  MX1 | -0.20869 [-0.50587 to 0.05456] | 2.03597 [0.85705 to 2.57300]
  NPC1L1 | 0.22706 [-0.03894 to 0.64205] | -0.14370 [-0.69620 to 0.04284]
  OAS1 | -0.16315 [-0.48203 to -0.02391] | 1.38768 [0.18495 to 1.52130]
  OAS2 | -0.07088 [-0.29292 to 0.08164] | 2.08119 [0.75112 to 2.30308]
  OAS3 | 0.05866 [-0.31366 to 0.19116] | 1.76892 [0.30701 to 2.17940]
  OASL | 1.03897 [0.61243 to 1.56387] | 2.27481 [2.04035 to 2.44387]
  PLSCR1 | -0.29797 [-0.38649 to -0.09644] | 0.63596 [0.46577 to 0.92180]
  PPARA | -0.51770 [-0.71264 to -0.12349] | -0.50756 [-0.84883 to -0.34797]
  PRKAB2 | 0.01071 [-0.20709 to 0.13838] | -0.30954 [-0.49940 to -0.17102]
  RSAD2 | -0.14051 [-0.43403 to 0.16345] | 1.60724 [0.24005 to 1.96854]
  STAT1 | 0.15195 [-0.07540 to 0.27268] | 1.44922 [0.72279 to 1.65143]
  TAP1 | 0.14096 [-0.06953 to 0.48128] | 0.68816 [-0.02488 to 1.01691]

2. Secondary Outcome: Rates of Rapid Virological Responder
Description: rapid virological response (HCV RNA <LLOQ Target not Detected) at week 4
Time Frame: Week 4 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 22 | 11

3. Secondary Outcome: Extended Rapid Virological Responder
Description: extended rapid virological response (HCV RNA <LLOQ Target not Detected at both weeks 4 and 12)
Time Frame: Both weeks 4 and 12 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 21 | 9

4. Secondary Outcome: End of Treatment Responder
Description: end of treatment response (HCV RNA <LLOQ Target not Detected at week24)
Time Frame: Week 24 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 20 | 8

5. Secondary Outcome: Sustained Virological Responder
Description: sustained virological response at follow-up week 12
Time Frame: Week 12 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 19 | 8

6. Secondary Outcome: Serum Aminotransferase Levels
Description: whether raw ALT value is in normal range which is less than 41 U/L.
Time Frame: Week 12 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 15 | 6

7. Secondary Outcome: Virological Relapse
Description: HCV RNA >= LLOQ level after therapy is stopped in a patient who previously achieved an end-of-treatment virological response
Time Frame: beyond Week 24 post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 1 | 0

8. Secondary Outcome: Rates of Asunaprevir and Daclatasvir Resistance
Time Frame: post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Number analyzed (Participants) | 22 | 13
Participants | 1 | 4

ADVERSE EVENTS:
Description: Two participants from genotype 1b arm were switched to genotype 1a.
Groups:
- Hepatitis C Virus Genotype 1A: Subjects will be started on combination therapy with asunaprevir, daclatasvir, peginterferon alfa-2a and ribavirin for 24 weeks.
  Asunaprevir, daclatsvir, peginterferon, ribavirin
- Hepatitis C Virus Genotype 1B: subjects will receive combination therapy with asunaprevir and daclatasvir alone for 24 weeks and undergo paired liver biopsies, pre-treatment and either at 2 or 4 weeks after starting therapy.
  Asunaprevir and Daclatsvir
Arm/Group | Hepatitis C Virus Genotype 1A | Hepatitis C Virus Genotype 1B
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/13
Other Adverse Events (participants affected / at risk) | 24/24 | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis C Virus Genotype 1A (N=24) | Hepatitis C Virus Genotype 1B (N=13)
Abdominal pain (Gastrointestinal disorders) | 14 (40) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 15 (90) | 12 (50)
Blurry vision (Eye disorders) | 10 (42) | 1 (1)
Buttock and leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Chest pain (Cardiac disorders) | 4 (4) | 1 (1)
Chest tightness (Cardiac disorders) | 2 (2) | 1 (1)
Chills (Infections and infestations) | 14 (58) | 4 (5)
Confusion (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (25) | 5 (18)
Coughing (Infections and infestations) | 3 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 14 (43) | 4 (12)
Dizziness (Nervous system disorders) | 9 (36) | 6 (21)
Drowsiness (General disorders) | 2 (3) | 0 (0)
Dry mouth (General disorders) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (132) | 7 (46)
Edema (Cardiac disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 24 (174) | 11 (88)
Fever (Infections and infestations) | 13 (30) | 3 (3)
Flu like sx (Infections and infestations) | 17 (82) | 6 (12)
Frequent urination (Renal and urinary disorders) | 17 (49) | 4 (13)
Hair loss (General disorders) | 13 (45) | 2 (10)
Headache (General disorders) | 20 (153) | 11 (39)
Insomnia (General disorders) | 10 (62) | 7 (26)
Irritability (General disorders) | 16 (80) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 17 (116) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 16 (89) | 1 (1)
Loose stool (Gastrointestinal disorders) | 2 (2) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 5 (5) | 0 (0)
Lump injection site (Product Issues) | 2 (2) | 0 (0)
Memory loss (General disorders) | 4 (4) | 0 (0)
Muscle aches (Musculoskeletal and connective tissue disorders) | 21 (138) | 2 (2)
Nasal stuffines (Infections and infestations) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (72) | 7 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nose bleeds (General disorders) | 2 (9) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 16 (62) | 0 (0)
Runny nose (Infections and infestations) | 3 (3) | 0 (0)
Shortness of breath (Cardiac disorders) | 17 (73) | 6 (18)
Sadness (Psychiatric disorders) | 8 (31) | 0 (0)
Shivers (Infections and infestations) | 2 (6) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Sore Throat (Infections and infestations) | 3 (3) | 1 (1)
Sore mouth (Infections and infestations) | 2 (3) | 0 (0)
Stomach cramps (Gastrointestinal disorders) | 11 (48) | 3 (8)
Sweating (Infections and infestations) | 2 (2) | 1 (1)
Tingling sensation (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (15) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
limb cramp (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Adrenaline (General disorders) | 0 (0) | 1 (1)
Bleeding from ear (General disorders) | 0 (0) | 1 (1)
Decreased sex drive (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ear drainage (Infections and infestations) | 0 (0) | 1 (1)
Equilibrium problems (Nervous system disorders) | 0 (0) | 1 (1)
Eye spots (Eye disorders) | 0 (0) | 1 (1)
Hand tremor (Nervous system disorders) | 0 (0) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Heavy legs (General disorders) | 0 (0) | 1 (1)
Hoarseness (Infections and infestations) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Lack of concentration (General disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Night Sweats (General disorders) | 0 (0) | 1 (4)
Nightmares (Psychiatric disorders) | 0 (0) | 1 (1)
Poor smell (General disorders) | 0 (0) | 1 (1)
Post BX shoulder pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Post BX site pain (Surgical and medical procedures) | 0 (0) | 1 (1)
R hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Right rib cage pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Stuffy nose (Infections and infestations) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Toe pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tooth abcess (Infections and infestations) | 0 (0) | 2 (2)
Tooth pain (Infections and infestations) | 0 (0) | 1 (1)
Warm (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes